CLINICAL TRIAL: NCT04212247
Title: Randomized Controlled Trial for Testing the Efficacy of Well-Being Therapy in Patients With Systemic Sclerosis
Brief Title: Trial on Outpatients With Systemic Sclerosis Treated With Well-Being Therapy or With a Control Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Fiammetta Cosci, Associate Professor in Clinical Psychology, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WBT in SSc
Record Dates: First submitted 2019-12-18; First posted 2019-12-26 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Systemic Sclerosis
Keywords: systemic sclerosis, well-being, psychological distress, suffering, mental pain, well-being therapy, psychotherapy
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: This is a pilot study, designed as a randomized (1:1) controlled trial, comparing WBT vs a control condition. The patients will receive a baseline assessment to confirm the diagnosis of systemic sclerosis, then socio-demographic information, information on pharmacological/non-pharmacological treatments, on the history of medical diseases and on the psychological status will be collected. Thereafter, the subjects will be randomly assigned to WBT or to a control condition. The subjects will be re-assessed at the end of session 4, 8 of treatment, and at 6-month follow-up.
Who Masked: Participant
Masking Description: Participants will not be informed if they will receive WBT or the control condition. At the end of the study they will receive this information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Well-being therapy (Experimental): WBT will be used as the only non-pharmacological therapeutic strategy and 8 sessions will be delivered every other week with a duration of 60 minutes each. The manualized WBT will be used (Fava, 2016). Thus, the initial phase will be concerned with self-observation of psychological well-being. Once the instances of well-being will be properly recognized, the patient will be encouraged to identify thoughts, beliefs, and behaviors leading to premature interruption of well-being (intermediate phase). The final part will involve cognitive restructuring of dysfunctional dimensions of psychological well-being and meeting the challenge that optimal experiences may entail.
  Interventions: Behavioral: Well-Being Therapy
- Control condition (Placebo Comparator): The control condition will include 8 every other week sessions based on Lifestyle and well-being National Institute for health and Care Excellence (NICE) guidelines (https://www.nice.org.uk/guidance/lifestyle-andwellbeing) and on World Health Organization 12 steps to healthy eating (http://www.euro.who.int/en/ health-topics/disease-prevention/nutrition/a-healthylifestyle). These sessions will inform participants about well-being and lifestyles which can influence it.
  Interventions: Behavioral: Control condition

INTERVENTIONS:
Behavioral: Well-Being Therapy — Well-Being Therapy (WBT) is a short-term psychotherapeutic strategy, that emphasizes self-observation with the use of a structured diary, interaction between patients and therapists and homework. WBT was based on the model of psychological well-being that was originally developed by Jahoda in 1958 and further refined by Ryff in 2014. The standard number of sessions is 8. The initial phase is concerned with self-observation of psychological well-being. Then, the patient is encouraged to identify thoughts, beliefs, and behaviors leading to premature interruption of wellbeing. The final part involves cognitive restructuring of dysfunctional dimensions of psychological well-being and meeting the challenge that optimal experiences may entail.
  Arms: Well-being therapy
Behavioral: Control condition — The control condition will include 8 sessions that will inform participants about well-being and lifestyles which can influence it. They will be articulated as follows. Session 1: illustrating the concept of lifestyle and well-being. Session 2 and session 3: illustrating healthy eating and steps to healthy eating. Session 4: illustrating physical exercise and how it promotes health. Session 5: illustrating smoking and tobacco and how they can damage health. Session 6: illustrating alcohol and how it can damage health. Session 7: illustrating drug misuse and how it can damage health. Session 8: illustrating sexual health. No access to specific WBT ingredients will be allowed.
  Arms: Control condition

SUMMARY:
Systemic sclerosis (SSc) is a rare and potentially life-threatening autoimmune disorder with a significant impact on health and quality of life. The non-pharmacological interventions address to psychological sequalae currently available are limited and have poor efficacy. Well-Being Therapy (WBT) is a brief psychotherapy which has shown efficacy in decreasing the relapse rates of depression in adults, in generalized anxiety disorder and in cyclothymia. WBT has never been tested in SSc and it might represent a useful complementary therapeutic option to improve SSc patients' well-being. The aim of the present study is to evaluate the psychological status of the SSc patients and to test the efficacy of WBT in a sample of SSc patients if compared to a control condition.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a rare, multisystem, chronic autoimmune connective tissue disease characterized by ﬁbrosis of the skin and internal organs, skin thickening, and decreased organ functioning leading to dermatologic, vascular, pulmonary, cardiac, gastrointestinal, neurological, musculoskeletal, and renal complications. SSc patients often suffer from psychological impairments, such as depression, anxiety about disease progression, body image dissatisfaction and low self-esteem. The non-pharmacological interventions for the treatment of the psychological sequelae of systemic sclerosis currently available are limited and have shown poor efficacy. Well-Being Therapy (WBT) is a brief psychotherapy which has been manualized in 2016 and has shown efficacy in randomized clinical trials. It showed to be effective in decreasing the relapse rates of depression in adults, it showed to be effective in generalized anxiety disorder and in cyclothymia. No psychological treatment aimed at empowering the level of psychological well-being rather than at working on distress in SSc patients have been implemented although it was shown that such kind of interventions directly increase the level of psychological well-being and indirectly decrease the level of psychological distress (i.e., anxious and depressive symptoms) in subjects affected by chronic diseases. The aim of the present study is to evaluate the psychological status of SSc patients with specific attention to suffering and mental pain, and to test the efficacy of WBT in SSc subjects if compared to a control condition. Thus, sixty outpatients with a diagnosis of SSc will be enrolled and will receive WBT or the control condition.

ELIGIBILITY:
Inclusion Criteria:

1. able and interested in participating to the research, as proved by signed Informed consent;
2. a diagnosis of SSc (limited or diffuse) according to LeRoy et al. (1998);
3. age higher than 18 years

Exclusion Criteria:

1. co-occurrence of psychiatric disorder(s) according to the Diagnostic and Statistical Manual of mental disorders, 5th edition (American Psychiatric Association, 2013) as diagnosed via the Mini-International Neuropsychiatric Interview;
2. currently under psychotherapy;
3. change of the pharmacological treatment (including psychotropic medications) during the last three months.
4. any other condition that, according to the Investigators' opinion, may alter the ability of the patient to follow study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Disability due to systemic sclerosis | change from baseline to 6-month follow up
  The primary outcome will be the level of disability due to systemic sclerosis, assessed via the Health Assessment Questionnaire Disability Index (minimum: 0, maximum: 40, the highest the score the highest the level of disability).

SECONDARY OUTCOMES:
Psychiatric status | change from baseline to 6-month follow up
  Psychiatric status assessed via the Mini-International Neuropsychiatric Interview (no score applicable)
Psychosomatic status | change from baseline to 6-month follow up
  Diagnostic Criteria for Psychosomatic Research-Revised Semi-Structured Interview (no score applicable)
Well-being | change from baseline to 6-month follow up
  World Health Organization-Five Well-Being Index (min: 0, max: 25, the highest score corresponds to the lowest level of well-being)
Psychological well-being | change from baseline to 6-month follow up
  the Psychological Well-Being Questionnaire (min: 0, max: 504, the highest score corresponds to the highest level of psychological well-being)
Euthymia | change from baseline to 6-month follow up
  Euthymia Scale (min: 0, max: 60, the highest score corresponds to highest level of euthymia)
Suffering | change from baseline to 6-month follow up
  Pictorial Representation of Illness and Self-Measure (min: 0, max: 30, the highest score corresponds to the lowest level of suffering)
Psychological distress | change from baseline to 6-month follow up
  Symptom Questionnaire (min: 0, max: 92, the highest score corresponds to the highest level of psychological distress)
Pain in the body | change from baseline to 6-month follow up
  Brief Pain Inventory (min: 0, max: 70, the highest score corresponds to highest level of pain)
Mental pain | change from baseline to 6-month follow up
  Mental Pain Questionnaire (min: 0, max: 20, the highest score corresponds to the highest level of mental pain)
Psychiatric symptoms | change from baseline to 6-month follow up
  Symptom Checklist-90-Revised (min: 0, max: 320, the highest score corresponds to the highest level of symptoms severity)
Harmony | change from baseline to 6-month follow up
  Visual analouge scale (min: 0, max: 100, the highest score corresponds to the highest level of harmony)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Rheumtoi Unit, Academic Hospital Careggi, Florence
  - Fiammetta Cosci, Florence

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Romanazzo S, Ceccatelli S, Mansueto G, Sera F, Guiducci S, Matucci Cerinic M, Cosci F. Well-Being Therapy in systemic sclerosis outpatients: a randomized controlled trial. Rheumatology (Oxford). 2025 Feb 1;64(2):667-674. doi: 10.1093/rheumatology/keae114. PMID 38366929